CLINICAL TRIAL: NCT02980536
Title: The Oncogenic Mutation Detection of Advanced NSCLC Patients by cSMART Liquid Biopsy and Dynamic Monitor of Tyrosine Kinase Inhibitor(TKI) Efficiency in Inner-Mongolia China
Brief Title: cSMART Liquid Biopsy and Dynamic Monitor of NSCLC Patients in Inner-Mongolia China
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Berry Genomics Co., Ltd. (Industry)
Collaborators: Shanghai Chest Hospital (Other); Baotou Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BerryGenomics NMB
Record Dates: First submitted 2016-11-27; First posted 2016-12-02 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Nonsmall Cell Lung Cancer; Adenocarcinoma
Keywords: NSCLC; TKI; Mutation; Liquid Biopsy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — There are two types of biospecimen collected in this study. One is the tumor tissue sample taken by biopsy. The other is the plasma sample from the blood.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate the mutation pattern of epidermal growth factor receptor (EGFR) and other TKI targeted gene during TKI treatment of advanced NSCLC patient with liquid biopsy.

DETAILED DESCRIPTION:
In the study, 200 advanced NSCLC patients will be recruited. All the patients will receive biopsy genotype assay and Circulating Single-Molecule Amplification and Resequencing Technology (cSMART) liquid biopsy. those patients who carry EGFR activating mutation and other TKI targeted activating mutation will receive TKI treatment. During the TKI treatment, every patients will take liquid biopsy assay to monitor the mutation status. the study will be ended when all the patients had a progressive disease (PD) in their targeted lesion

ELIGIBILITY:
Inclusion Criteria:

* NSCLC adenocarcinoma patients confirmed by pathologist
* Initial, non-operative patients with stage III & IV adenocarcinoma
* Older than 18 years old
* Subjects have no major organ dysfunction. In detail, Liver Function: TBiL≤1.5 ULN ( Upper Limit of Normal); Serum GPT (Glutamate-Pyruvate Transaminase ):≤2 ULN, Renal Function: ScR≤1.2 ULN; BUN≤1.2 ULN, BM (Bone Marrow) Reserve: WBC (White Blood cell Count) ≥4.0×e9/L; ANC≥2.0×e9/L，PLT≥100×e9/L，HGB≥100g/L.

PS (Performance Status) Score: less than 2, Expected Survival Time: More than 3 months;

* Have a clear measurable tumor lesion in lung,under RIEST.
* Without severe drug allergy
* Patients participate in this trail must sign the informed consent

Exclusion Criteria:

* Patients with brain metases related syndrome
* Patients with bone metases related complication
* Patients with cognitive disorder
* Patients with major organ dysfunction and severe cardiopathy include congestive heart-failure, uncontrolled arrhythmia, angina with long term treatment, VHD (Valvular Heart Disease), myocardial infraction, RHTN (Resistant Hypertension).
* Patients with other severe complication and excluded by the researcher.
* Patients who are allergy with the TKI in this trail.
* Patients who participated in other trails or with anti-tumor treatments
* Patients who receive radiotherapy at the site of curative effect observation
* Patients who receive allogenic blood transfusion within 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Stage III and Stage IV NSCLC, adenocarcinoma.
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The TKI resistance gene mutation pattern in plasma DNA of TKI treated patient | 1.5 years
  The researcher would like to find out the change of mutation in plasma DNA of the patients who received TKI treatment by a liquid biopsy method.

SECONDARY OUTCOMES:
The concordance of gene mutation pattern between liquid biopsy and traditional cancer tissue biopsy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shun Lu, MD/PhD, Study Chair — Shanghai Chest Hospital
Locations (9):
- China (9):
  - Baogang Hospital, Baotou, Inner Mongolia
  - Baotou Cancer Hospital, Baotou, Inner Mongolia
  - Northern Hospital Baotou, Baotou, Inner Mongolia
  - Baotou Centry Hospital, Baotou, Inner Mongolia
  - Bayan Nur Hospital, Bayan Nur, Inner Mongolia
  - The Inner Mongolia Autonomous Region Cancer Hospital, Hohhot, Inner Mongolia
  - The Inner Mongolia Autonomous Region People's Hospital, Hohhot, Inner Mongolia
  - The First Affiliated Hospital of Inner Monglia Medical University, Hohhot, Inner Mongolia
  - Dalad Banner People's Hospital, Ordos, Inner Mongolia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Z, Cheng G, Han X, Mu X, Zhang Y, Cui D, Liu C, Zhang L, Fan Z, Ma L, Yang L, Di J, Cram DS, Shi Y, Liu D. Application of Single-Molecule Amplification and Resequencing Technology for Broad Surveillance of Plasma Mutations in Patients with Advanced Lung Adenocarcinoma. J Mol Diagn. 2017 Jan;19(1):169-181. doi: 10.1016/j.jmoldx.2016.09.008. Epub 2016 Nov 19. PMID 27870944
- [Background] Chai X, Ren P, Wei B, Ma J, Mai L, Cram DS, Song Y, Guo Y. A comparative study of EGFR oncogenic mutations in matching tissue and plasma samples from patients with advanced non-small cell lung carcinoma. Clin Chim Acta. 2016 Jun 1;457:106-11. doi: 10.1016/j.cca.2016.04.003. Epub 2016 Apr 9. PMID 27071701
- [Background] Song Y, Zhou X, Huang S, Li X, Qi Q, Jiang Y, Liu Y, Ma C, Li Z, Xu M, Cram DS, Liu J. Quantitation of fetal DNA fraction in maternal plasma using circulating single molecule amplification and re-sequencing technology (cSMART). Clin Chim Acta. 2016 May 1;456:151-156. doi: 10.1016/j.cca.2016.03.005. Epub 2016 Mar 15. PMID 26993877
- [Background] Lv W, Wei X, Guo R, Liu Q, Zheng Y, Chang J, Bai T, Li H, Zhang J, Song Z, Cram DS, Liang D, Wu L. Noninvasive prenatal testing for Wilson disease by use of circulating single-molecule amplification and resequencing technology (cSMART). Clin Chem. 2015 Jan;61(1):172-81. doi: 10.1373/clinchem.2014.229328. Epub 2014 Nov 6. PMID 25376582